Date: 1 March 2020

**Study Name:** Comparison Of The Incidence Of Recurrent Laryngeal Injury Following The Dissection Of The Nerve By Cranio-Caudal And Lateral Approach By Using Introperative Nerve Monitoring

Statistical Analysis Plan: The Statistical Package for Social Sciences (SPSS) for Windows Version 21.0 (Armonk, NY: IBM Corp.) was used for statistical analysis. The continuous variables are summarised as mean  $\pm$  standard deviation. The differences between the groups were assessed using the Student's t-test and a Mann-Whitney U test for normally distributed and non-normally distributed data, respectively. Univariate analysis by Chi-square test was performed to test differences in proportions. Statistically significant results obtained from the univariate analysis were subjected to multivariate logistic regression. A p value <0.05 was considered to be statistically significant.